CLINICAL TRIAL: NCT01751620
Title: Project ACCEPT: Engaging Newly Diagnosed HIV+ Youth in Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATN 108
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-10

CONDITIONS: HIV Positive Youth That Are Newly Engaged in Care
MeSH Terms: interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project ACCEPT (Experimental): Participants randomized to the intervention (Project ACCEPT) arm.
  Interventions: Behavioral: Project ACCEPT
- HEALTH (Active Comparator): Participants randomized to the comparison (HEALTH) arm.
  Interventions: Behavioral: HEALTH

INTERVENTIONS:
Behavioral: Project ACCEPT — The intervention, Project ACCEPT, combines weekly individual and group sessions that address a range of issues that impact engagement in care for youth living with HIV, including stigma, disclosure, health relationships, substance use, and future life plans.
  Other Names: Adolescents Coping, Connecting, Empowering and Protecting Together
  Arms: Project ACCEPT
Behavioral: HEALTH — The comparison condition, HEALTH, matches Project ACCEPT in number of sessions and duration. The weekly sessions will cover information on alcohol, drugs, HIV and other sexually transmitted diseases (STDs) to meet the ethical responsibility to provide risk reduction information to youth assigned.
  Arms: HEALTH

SUMMARY:
The proposed study is a two-group randomized repeated measures design that will examine the efficacy of Project ACCEPT (Adolescents Coping, Connecting, Empowering and Protecting Together) to improve engagement in care among youth newly diagnosed with HIV at five AMTU sites across the United States. Youth will be randomized into one of two study arms; Project ACCEPT, the intervention, or HEALTH, the health education attention-controlled comparison condition. Both arms consist of two individual sessions followed by six group sessions and a final individual session which is expected to take approximately nine weeks after which youth will have four follow-up visits at the following time points:

* post intervention (immediately after the last session);
* 3 months post the last session;
* 6 months post the last session; and
* 12 months post the last session. The trial will be repeated in up to three waves.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected and aware of his/her status as documented by medical record review or verbal verification by provider (i.e., medical or mental health care provider, case manager, social worker, etc.);
* Received HIV diagnosis within the past 12 months (+ 3 months) at the time of consent/assent as documented by medical record review or verbal verification with referring professional (i.e., medical or mental health care provider, case manager, social worker, etc.);
* Between the ages of 16-24 (inclusive) at the time of informed consent/assent;
* Receives services at one of the selected AMTUs or one of their community partners;
* Willing to participate in both the individual and group sessions;
* Ability to speak and understand spoken English;
* Able to understand and willing to provide signed informed consent/assent in English or Spanish; and
* Willingness to provide signed informed consent or assent with parental/legal guardian permission as applicable.

Exclusion Criteria:

* Participated in a previous wave, if enrolling into Wave 2 or 3;
* Intoxicated or under the influence of alcohol or other substances at the time of consent/assent;
* Visibly distraught and/or visibly emotionally unstable (i.e., exhibiting suicidal, homicidal, or violent behavior) in the opinion of the site personnel would interfere with the ability to give true informed consent; and
* Any concurrent participation in other behavioral studies. Permission from the protocol team may be provided for uncertain cases.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 167 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Examine the efficacy of Project ACCEPT compared with an attention-controlled health education comparison intervention | 3 years
  Conduct a randomized controlled trial to examine the efficacy of Project ACCEPT compared with an attention-controlled health education comparison intervention (HEALTH). The goals of the intervention are to improve engagement in care, decrease psychosocial barriers to care, and decrease sexual risk for youth newly diagnosed with HIV.

SECONDARY OUTCOMES:
Explore the relationship between HIV biomarkers and participant's level of engagement in care | 3 years
  Explore the relationship between HIV biomarkers (i.e., CD4 and viral load) and participant's level of engagement in care.

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Study Chair — Adolescent Trials Network; Gary Harper, PhD, Study Chair — Adolescent Trials Network
Locations (4):
- United States (4):
  - University of Miami School of Medicine, Miami, Florida
  - Stroger Hospital and the CORE Center, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - St. Jude Childrens Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: ATN website — http://www.atnonline.org